CLINICAL TRIAL: NCT06511960
Title: Impact of Four Weeks of Astaxanthin Supplementation at Varied Doses on Muscle Pain, Muscle Damage Markers, and Total Antioxidant Status in Exercising Males: A Randomized Controlled Trial
Brief Title: Effects of Astaxanthin Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Muhammed Mustafa Atakan, Associate Professor of Exercise Physiology, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: IMU-GETAT-E-95961207
Record Dates: First submitted 2024-07-09; First posted 2024-07-22 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Dietary Supplements
Keywords: Astaxanthin; supplements; antioxidant; muscle damage; resistance exercise
MeSH Terms: interventions — astaxanthine; Methods

STUDY DESIGN:
Intervention Model Description: Placebo-controlled, double-blind and three-group parallel design
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Astaxanthin (12 mg/day) group (Active Comparator): In this group, participants ingested either 12 mg/day (AX12) for 4 weeks.
  Interventions: Other: Astaxanthin (12 mg/day) intervention
- Astaxanthin (36 mg/day) group (Active Comparator): In this group, participants ingested either 36 mg/day (AX36) for 4 weeks.
  Interventions: Other: 36 mg/day astaxanthin intervention
- Placebo (Placebo Comparator): In this group, participants ingested the placebo capsules that were identical in appearance and dimensions to the astaxanthin supplement.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Astaxanthin (12 mg/day) intervention — 12 mg/day astaxanthin was administrated to all participants in the astaxanthin 12 mg/day groupfor 4 weeks. Following this supplementation protocol, we assessed the muscle damage markers (creatine kinase and lactate dehydrogenase), total antioxidant status (malondialdehyde and uric acid), and muscle pain levels were evaluated using the Numerical Visual Pain Scale0-10.
  Arms: Astaxanthin (12 mg/day) group
Other: 36 mg/day astaxanthin intervention — 36 mg/day astaxanthin was administrated to all participants in the astaxanthin 36 mg/day group for 4 weeks. Following this supplementation protocol, we assessed the muscle damage markers (creatine kinase and lactate dehydrogenase), total antioxidant status (malondialdehyde and uric acid), and muscle pain levels were evaluated using the Numerical Visual Pain Scale0-10.
  Arms: Astaxanthin (36 mg/day) group
Other: Placebo — 12 mg/day placebo was administrated to all participants in the placebo group for 4 weeks. Following the placebo supplementation, we assessed the muscle damage markers (creatine kinase and lactate dehydrogenase), total antioxidant status (malondialdehyde and uric acid), and muscle pain levels were evaluated using the Numerical Visual Pain Scale0-10.
  Arms: Placebo

SUMMARY:
Astaxanthin is a potent antioxidant and anti-inflammatory carotenoid. Research examining whether astaxanthin (AX) could counteract exercise-induced muscle damage and improve exercise capacity reported inconsistent results.Therefore, the aim of this study was to explore the impact of 4 weeks supplementation with AX on muscle damage markers, total antioxidant status, and subjective marker of muscle pain. Twenty-four males were randomly assigned to the AX12 group (12 mg/day; n=8), AX36 group (36 mg/day; n=9), or placebo group (PLC; n=7). After 4 weeks of supplementation, blood samples were collected at rest, immediately after, and at 2, 24, 48, and 72 hours following eccentric arm exercise at 85% of predetermined one repetition maximum to assess muscle damage markers (creatine kinase and lactate dehydrogenase), total antioxidant status (malondialdehyde and uric acid), and muscle pain levels were evaluated using the Numerical Visual Pain Scale0-10.

DETAILED DESCRIPTION:
This study followed a placebo-controlled, double-blind (participants and co-researcher administering the supplementation), and three-group parallel design to examine the effects of an AX supplement on muscle pain, muscle damage markers, and total antioxidant status (TAS).

Participants reported to the laboratory on 2 separate occasions: one initial session to measure anthropometrics and 1-repetition maximum (1RM) strength of the arm muscles and as well as to collect resting venous blood samples, prior to the four-week supplementation period. Upon arrival at the laboratory for their initial visits, each participant underwent measurements of body mass (MC 780 ST Black) and body height (Telescopic Height Meter), after which resting venous blood samples were collected from the median antecubital vein by a healthcare professional.

Following these baseline measurements, participants were assigned to one of the groups through a strict randomization process, which included selecting boxes numbered up to 24, all with the same size, color, and pattern. Participants were asked to choose one of the random numbers accompanied by an independent person other than the researchers. This process was recorded by the supervisor in paper-based surveys and digitally. Subsequently, all participants were instructed to consume their corresponding supplements (4 mg/day AX, 12 mg/day AX or 12 mg/day PLC) for 4 weeks.

After the 4 weeks of supplementation, participants reported to the laboratory for the post-supplementation measurements that included the collection of blood samples at rest, immediately after, as well as at 2, 24, 48, and 72 hours following completing eccentric arm exercises performed at 85% of predetermined 1RM.

Before obtaining blood samples (i.e., immediately after, and at 2, 24, 48, and 72 hours after exercises), participants were asked to assess their current pain levels using the Numerical Visual Pain Scale (NRS, ranging between 0-10 and 0-100) to determine any correspondence with muscle damage markers in the blood 25.

All participants were instructed to abstain from taking any medications for a minimum of 7 days prior to the study and to avoid consuming vitamins, foods, or supplements containing antioxidants, as well as analgesics, aspirin, or any other anti-inflammatory drugs throughout the duration of the study. A list of AX-rich foods, beverages and vitamins was provided to each participant prior to testing and all participants were asked to avoid these items during both 4-week supplementation periods and to maintain their regular eating habits and refrain from strenuous exercise to minimize the risk of muscle damage. A WhatsApp group was created for the purpose of monitoring the participants' supplement use.

To ascertain the extent of product usage, a survey form created using Google Forms was disseminated during the supplementation period. Participants were required to approve the form on a daily basis. At the end of each day, the data entered into the Excel file created using OneDrive was reviewed by at least one researcher.

ELIGIBILITY:
Inclusion Criteria:

Healthy males engaging in recreational activity Aged between 20 and 30 years Non-smoker Not participating in any structured training regimen (i.e., endurance or resistance training programs)

Exclusion Criteria:

Use of any supplement or regular medications, Having hypothyroidism or hyperthyroidism.

Ages: 19 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-04-15 (Actual)

PRIMARY OUTCOMES:
Assessment of Muscle Pain | 2-6 months
  The pain sensation in the participants' elbow extensor and elbow flexor muscles was assessed using the NRS. NRS is one of the most widely used scales due to its simplicity and effectiveness for assessing pain intensity across various medical settings and research studies. This scale rates individuals' pain on a scale from 0 to 10, with 0 representing no pain and 10 representing the worst pain imaginable (1-3: mild pain, 4-6: moderate pain, 7-10: severe pain). In this study, we evaluated the participants' pain immediately after exercise and at 2, 24, 48, and 72 hours post-exercise. For this, participants were instructed to move their arms, which were used in the 1RM eccentric arm exercise, from a fully bent position to a fully straight position. During this movement, participants were asked to rate the intensity of pain they experienced.
Assessment of Malondialdehyde (MDA) | 2-6 months
  MDA is a natural product of lipid peroxidation. Lipid peroxidation is a well-known mechanism of animal and plant cell damage and suggests the level of oxidative stress or damage in cells and tissues. The MDA levels were assessed using thiobarbituric acid reactive substances assay kits (Cayman TBARS, Cayman Chemical, Ann Arbor, Michigan, USA, item no. 10009055) based on the trichloroacetic acid method in accordance with the manufacturer's instructions. The absorbance measurements were taken using the ChemWell 2910 ELISA reader device (Awareness, Technology, Inc. Martin Hwy. Palm City, USA). The results were presented as mmol Trolox Equiv./L for TAS and µM for MDA.
Assessment of Total Antioxidant Status (TAS) | 2-6 months
  Serum TAS (mmol Trolox Equiv./L) was determined using the Rel Assay Diagnostics kit (Mega Tip, Gaziantep, Turkey) using the method developed by Erel. This method mediates the production of a hydroxyl radical. The hydroxyl radical is the most powerful among biological radicals. In the test, the Fe ion solution present in reagent 1 is mixed with hydrogen peroxide present in reagent 2. Using this method, the antioxidative effect of the sample against the strong free radical reactions initiated by the hydroxyl radical produced was measured. The test had excellent sensitivity values of > 97%. Results were expressed as millimoles of Trolox equivalents per liter (mmol Trolox Equiv./L).
Assessment of Muscle Damage Markers: Creatine kinase (CK) and Lactate Dehydrogenase (LDH) | 2-6 months
  Serum CK and LDH were analyzed on a fully automatic analyzer (Roche Cobas Integra 400 Plus, Roche Diagnostics GmbH, Mannheim, Germany) using ROCHE kits (Mannheim, Germany). Data were calculated using linear regression and measurements were taken at 550 nm.
Assessment of Uric Acid | 2-6 months
  Uric acid were analyzed on a fully automatic analyzer (Roche Cobas Integra 400 Plus, Roche Diagnostics GmbH, Mannheim, Germany) using ROCHE kits (Mannheim, Germany). Data were calculated using linear regression and measurements were taken at 550 nm.

SECONDARY OUTCOMES:
Measurement of One-Repetition Maximum (1RM) Arm Strength | 1-5 months
  The 1RM arm strength of participants was quantified by measuring the number of biceps curl repetitions performed in a seated position, following a 10-repetition warm-up set with a load equivalent to 50% of the estimated 1RM based on the participants' experience. Following a one-minute recovery period, a first set of five repetitions was performed at 75% of 1RM. After a two-minute recovery period, a second set of three repetitions was performed at approximately 90% of 1RM. Finally, after a 4-minute recovery, incremental increases of 2.5 kg were applied for each subsequent 1RM attempt until failure. After 4 weeks of supplementation, all participants performed an eccentric arm exercise of 10 sets × 10 repetitions at 85% of 1RM, with 3-minute passive rest intervals between each set, following a 10-repetition warm-up with 50% of 1RM.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammed Atakan, PhD, Principal Investigator — Hacettepe University
Locations (1):
- Muhammed Atakan, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Howatson G, van Someren KA. The prevention and treatment of exercise-induced muscle damage. Sports Med. 2008;38(6):483-503. doi: 10.2165/00007256-200838060-00004. PMID 18489195
- [Background] Markus I, Constantini K, Hoffman JR, Bartolomei S, Gepner Y. Exercise-induced muscle damage: mechanism, assessment and nutritional factors to accelerate recovery. Eur J Appl Physiol. 2021 Apr;121(4):969-992. doi: 10.1007/s00421-020-04566-4. Epub 2021 Jan 8. PMID 33420603
- [Background] Bloomer RJ. The role of nutritional supplements in the prevention and treatment of resistance exercise-induced skeletal muscle injury. Sports Med. 2007;37(6):519-32. doi: 10.2165/00007256-200737060-00005. PMID 17503877
- [Background] McArdle A, Vasilaki A, Jackson M. Exercise and skeletal muscle ageing: cellular and molecular mechanisms. Ageing Res Rev. 2002 Feb;1(1):79-93. doi: 10.1016/s0047-6374(01)00368-2. PMID 12039450
- [Background] Vina J, Gomez-Cabrera MC, Lloret A, Marquez R, Minana JB, Pallardo FV, Sastre J. Free radicals in exhaustive physical exercise: mechanism of production, and protection by antioxidants. IUBMB Life. 2000 Oct-Nov;50(4-5):271-7. doi: 10.1080/713803729. PMID 11327321
- [Background] He F, Li J, Liu Z, Chuang CC, Yang W, Zuo L. Redox Mechanism of Reactive Oxygen Species in Exercise. Front Physiol. 2016 Nov 7;7:486. doi: 10.3389/fphys.2016.00486. eCollection 2016. PMID 27872595
- [Background] Kuru D, Aktitiz S, Atakan MM, Kose MG, Turnagol HH, Kosar SN. Effect of Pre-exercise Sodium Citrate Ingestion on Repeated Sprint Performance in Soccer Players. J Strength Cond Res. 2024 Mar 1;38(3):556-562. doi: 10.1519/JSC.0000000000004651. Epub 2024 Jan 19. PMID 38241467
- [Background] Bongiovanni T, Genovesi F, Nemmer M, Carling C, Alberti G, Howatson G. Nutritional interventions for reducing the signs and symptoms of exercise-induced muscle damage and accelerate recovery in athletes: current knowledge, practical application and future perspectives. Eur J Appl Physiol. 2020 Sep;120(9):1965-1996. doi: 10.1007/s00421-020-04432-3. Epub 2020 Jul 13. PMID 32661771
- [Background] Brotosudarmo THP, Limantara L, Setiyono E, Heriyanto. Structures of Astaxanthin and Their Consequences for Therapeutic Application. Int J Food Sci. 2020 Jul 20;2020:2156582. doi: 10.1155/2020/2156582. eCollection 2020. PMID 32775406
- [Background] Higuera-Ciapara I, Felix-Valenzuela L, Goycoolea FM. Astaxanthin: a review of its chemistry and applications. Crit Rev Food Sci Nutr. 2006;46(2):185-96. doi: 10.1080/10408690590957188. PMID 16431409
- [Background] Cao Y, Yang L, Qiao X, Xue C, Xu J. Dietary astaxanthin: an excellent carotenoid with multiple health benefits. Crit Rev Food Sci Nutr. 2023;63(18):3019-3045. doi: 10.1080/10408398.2021.1983766. Epub 2021 Sep 28. PMID 34581210
- [Background] Brown DR, Gough LA, Deb SK, Sparks SA, McNaughton LR. Astaxanthin in Exercise Metabolism, Performance and Recovery: A Review. Front Nutr. 2018 Jan 18;4:76. doi: 10.3389/fnut.2017.00076. eCollection 2017. PMID 29404334
- [Background] Waldman HS, Bryant AR, Parten AL, Grozier CD, McAllister MJ. Astaxanthin Supplementation Does Not Affect Markers of Muscle Damage or Inflammation After an Exercise-Induced Muscle Damage Protocol in Resistance-Trained Males. J Strength Cond Res. 2023 Jul 1;37(7):e413-e421. doi: 10.1519/JSC.0000000000004408. Epub 2023 Jan 18. PMID 36727984
- [Background] Naguib YM. Antioxidant activities of astaxanthin and related carotenoids. J Agric Food Chem. 2000 Apr;48(4):1150-4. doi: 10.1021/jf991106k. PMID 10775364